CLINICAL TRIAL: NCT03089489
Title: Role of Lung Surfactant Proteins in Donor Lung to Predict Primary Graft Dysfunction in Lung Recipients
Brief Title: Lung PGD Biomarkers in Organ Donors
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital of Mont-Godinne (Other)
Responsible Party: Principal Investigator, Asmae Belhaj, MD, PhD, University Hospital of Mont-Godinne
Other Study IDs: B039201731131
Record Dates: First submitted 2017-03-07; First posted 2017-03-24 (Actual); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Lung Transplant Failure
Keywords: Primary graft dysfunction; Lung transplantation; Surfactant Protein; inflammation
MeSH Terms: conditions — Primary Graft Dysfunction; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Lung and blood samples in organ donors
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lung recipients with PGD: in the first 72 hours following lung transplantation, the lung recipients have blood gases and chest X-Ray to assess the occurrence of primary graft dysfunction. Chest X-Ray infiltrate and pathological PaO2/FiO2 ratio describe PGD occurence
  Interventions: Diagnostic Test: lung biomarkers in organ donor for PGD in lung recipient
- Lung recipients PGD Free: In the first 72 hoours following lung transplantation, if the Cest X-ray is normal, the patient is considered PGD-free
  Interventions: Diagnostic Test: lung biomarkers in organ donor for PGD in lung recipient

INTERVENTIONS:
Diagnostic Test: lung biomarkers in organ donor for PGD in lung recipient — Lung biopsies in organ donor before and after cold ischemia

SUMMARY:
PGD is a syndrome characterized by alveolocapillary barrier structural and functional alterations with surfactant inactivation and vascular permeability increase, which cause lung edema, parenchymal infiltrate and progressive hypoxemia.

PGD may be enhanced in lung donor. Inflammatory and structural changes may be present in the lungs before organ recovery and/or after organ preservation. The investigators aim to identify the surfactant protein, inflammatory and structural changes in lung donor before and after cold ischemia, and biomarkers to PGD in lung recipients.

DETAILED DESCRIPTION:
Primary graft dysfunction (PGD) is responsible of high early mortality in lung transplanted patients.

Rationale

The evolution of lung transplantation may be complicated by primary graft dysfunction (PGD), a form of acute respiratory distress syndrome caused by ischemia-reperfusion-related phenomena. PGD occurs in 15-50% of cases and is responsible for a significant increase in mortality, duration of assisted ventilation and length of stay in intensive care. It is also an important risk factor for the medium-term development of acute and long-term rejection, of bronchiolitis obliterans syndrome (BOS) - chronic rejection - which drastically reduces the survival of the graft.

Surfactant proteins comprising the secretory protein of Clara cells (16-kd Clara cell protein-CC16) and surfactant proteins -A (SP-A), -B (SP-B) and -D (SP- D) are recognized as markers of the permeability of the alveolocapillary barrier.

Based on these findings, we postulate that the gene expression of CC16, SP-A, -B and D is altered in pulmonary biopsies performed in donors of patients developing primary graft dysfunction after pulmonary transplantation compared to those performed in the donors of patients free of this syndrome.

This study could therefore be a complementary means of objective assessment of lung quality prior to transplantation.

Aims and Objectives

1. Describe, in the organ donor, changes in expression of Clara Cell Protein (CC16), surfactant-associated proteins (A, B or D), pro- and anti-inflammatory cytokines in circulating blood and lung tissue during organ recovery.
2. Describe the biological and structural changes after the period of cold ischemia.
3. Establish a correlation between biomarkers in the organ donor and the occurrence of acute graft dysfunction in the lung recipient.

Material and method

Inclusion Criteria

All lung organ donor patients referred to our network and their recipients will be included after obtaining their informed consent.

Data Collection

In the donor, we will record demographic data (age, sex), history, cause of death, blood gas measurement, chest x-ray protocol, blood biological parameters, duration of brain death if appropriate and hot ischemia time if appropriate and protocol of bacteriological analyzes.

In the recipient, we will record the demographic data (age, sex), indication of transplantation, results of right catheterization performed on pre-transplantation, standard intraoperative data, immunosuppression, Blood gas, chest x-ray protocol, filling balance and blood biological parameters at 24, 48 and 72h. The declamping times are recorded.

Patients are automatically followed up for the rest of their lives. Iterative biopsies are performed in the first year to detect possible acute rejection. The data will be included in our study.

Biological samples

In the donor, before the perfusion of the preservation solutions, 18 cc of peripheral blood are taken (dry tube, 9 cc). 1 tube will be stored at -80 ° C., the other will be centrifuged (15 minutes, 10000 / min, 20 ° C.) and then the serum will be stored at -80 ° C.

Immediately after lung recovery, a pulmonary biopsy (6 cm2) is performed at the lower lobes.

A fragment will be immediately placed in liquid nitrogen and stored at -80 ° C. A second fragment is stored in formalin for 24h and then stored in paraffin blocks.

Before implantation, at the end of the preservation period, a new lung biopsy is performed in the lower lobes.

Biological analyzes

Histological examination and gradation

Lung tissues fixed in formalin are stained with hematoxylin-eosin to gradate lung lesions [(1) neutrophil infiltration, (2) airway epithelial cell damage, (3) interstitial edema, (4) Hyaline membrane and (5) hemorrhage].

Inflammation, apoptosis and Surfactant proteins

O Tissue mRNA measurements: in real time Quantification PCR (RTQ-PCR)

O Tissue peptide measurements: Western Blot - ELISA - MILLIPLEX

O Treatment of blood samples and analyzes: ELISA - MILLIPLEX

Protein inflammatory cytokines (TNF-alpha, IL-6, IL-8, IL-1, IL33) (IL-10), intercellular adhesion molecules (ICAM-1, VCAM-1), apoptosis (Bax, Bcl2, Caspases)

Evaluation of apoptosis: TUNEL - Immunohistochemistry

ELIGIBILITY:
Inclusion Criteria:

* All organ donors and their lung recipients who reached the criteria for lung recovery and transplantation

Exclusion Criteria:

* None

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All lung donors and their lung recipients who reached the criteria for lung recovery and transplantation
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-04-01 (Estimated); Primary Completion 2022-03-08 (Estimated); Study Completion 2024-03-08 (Estimated)

PRIMARY OUTCOMES:
Lung Biomarkers for primary graft dysfunction in organ donors | 5-7 years
  The investigators aim te describe lung donor structural and molecular changes in relation of PGD occurrence in recipient.

CONTACTS AND LOCATIONS:
Overall Officials: Asmae Belhaj, MD, PhD, Principal Investigator — CHU UCL Namur

IPD SHARING:
Plan to Share IPD: No